CLINICAL TRIAL: NCT01063426
Title: Reload of High Dose Atorvastatin for Preventing Deep Vein Thrombosis in Statin Users Undergoing Total Knee Replacement Arthroplasty: RE-STOP-DVT Study- A Prospective Randomized Controlled Trial
Brief Title: Re-STOP DVT: Reload of High Dose Atorvastatin for Preventing Deep Vein Thrombosis in Statin Users
Acronym: Re-STOP DVT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Hallym University Medical Center, Hallym University Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009-I055
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2010-02

CONDITIONS: Thrombosis; Prevention; Surgery
Keywords: Statin; Vein
MeSH Terms: conditions — Thrombosis | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin + enoxaparine arm (Experimental): High dose atorvastatin arm before index surgery+ conventional enoxaparin
  Interventions: Drug: High dose Atorvastatin+enoxaparin
- Conventional Enoxaprin (Active Comparator): Conventional Enoxaparin before 12hr and on 1-7th day after index surgery
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: High dose Atorvastatin+enoxaparin — High dose atorvastatin 80mg/day for 7days after index surgery (total knee replacement arthroplasty, TKRA). At the same time Enoxaparin 40mg SQ/day 12hr before TKRA and from 1day to 7day after TKRA should be administered.
  Arms: Atorvastatin + enoxaparine arm
Drug: Enoxaparin — Enoxaparin 40mg SQ/day 12hr before TKRA and on day 1 to day7 after TKRA should be administered.
  Arms: Conventional Enoxaprin

SUMMARY:
Reload of high dose statin may have potential for preventing deep vein thrombosis (DVT) in patients on statin undergoing total knee replacement arthroplasty.

A body of evidence have been reported that reloading of atorvastatin have efficacy in reducing periprocedural myocardial infarction and contrast induced nephropathy. These effects are considered to be mainly due to their antioxidant anti-thrombotic and anti-inflammatory property.

We, therefore, hypothesize that high dose atorvastatin re-loading may prevent DVT.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are going to receive total knee replacement arthroplasty from any cause.
* < 19 years old

Exclusion Criteria:

* patients with cancer
* Patients receiving anticoagulant agents from any cause
* current statin users
* expecting survival from other co-morbidity < 1year
* Bed ridden patient
* AST, ALT > 3times of upper normal limit
* CK> upper normal limit
* pregnancy
* patients who receives hormone replacement therapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Development of deep vein thrombosis diagnosed and confirmed by CT angiography at lower extremities | 7days after index surgery

SECONDARY OUTCOMES:
D-dimer, lipid panel (Total cholesterol, TG, HDL, LDL), hsCRP, CK, transaminase, ALP | 7days, 1month, 2month after index surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Ho Jo, MD, Principal Investigator — Hallym University Medical Center; Sang-Ho Jo, MD, Study Chair — Hallym University Medical Center
Locations (1):
- Hallym University Sacred Heart Hospital, Department of Cardiology and Orthopedic Surgery, Anyang-si, Gyeonggi-do, South Korea